CLINICAL TRIAL: NCT05520944
Title: Accelerating COVID-19 Clinical Recovery in the Outpatient Setting: Retrospective Data Collection and Analysis of COVID-19 Patients Treated With ClorNovir® (Chlorpheniramine Maleate (0.4% Nasal Spray)
Brief Title: Accelerating COVID-19 Clinical Recovery in the Outpatient Setting: Retrospective Analysis
Acronym: ACCROS-R
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Ferrer BioPharma (Industry)
Collaborators: Clinica Union Medica Del Norte, S.A.S., Santiago, República Dominicana (Unknown)
Responsible Party: Sponsor
Other Study IDs: DFB-004
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; COVID-19 Pandemic; COVID-19 Respiratory Infection; SARS CoV 2 Infection; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19 | interventions — Chlorpheniramine; Nasal Sprays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Retrospective Data Collection
  Interventions: Drug: ClorNovir® (Chlorpheniramine) 0.4% Nasal Spray

INTERVENTIONS:
Drug: ClorNovir® (Chlorpheniramine) 0.4% Nasal Spray — Patients will have received treatment with ClorNovir® as prescribed by their physician at the approved dose per local prescribing information, as part of their COVID-19 clinical recovery.
  Other Names: Chlorpheniramine Nasal Spray; ClorNovir®

SUMMARY:
The purpose of this retrospective study is to evaluate the effectiveness of CPM nasal spray as part of the treatment of COVID-19 and its impact on clinical symptoms. Two cohort groups will be compared (CPM vs. standard care). The hypothesis to be tested is that patients treated with CPM nasal spray showed more rapid clinical improvement than those treated with standard of care alone. Clinical improvement will be evaluated by the total number of days with the manifestation of COVID-19 symptoms, including cough, nasal congestion, ageusia, and anosmia, among others. The rate of hospitalization between the cohorts will also be evaluated.

DETAILED DESCRIPTION:
The following are categories of interest in patients with COVID-19 treated with ClorNovir:

* Clinical outcomes, as assessed by clinical assessments of clinical symptoms, and incidence of significant clinical events
* Clinical recovery, as assessed by patient-reported outcome measures and clinician-reported outcomes.

The safety objective is to assess the safety and tolerability of ClorNovir.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a documented diagnosis of SAR-CoV-2
* Patients with positive RT-PCR or antigen test for SARS-CoV-2 in nasopharyngeal or oropharyngeal swabs
* Both vaccinated and unvaccinated (high-risk) persons will be included.
* Willing and able to provide written informed consent (ages greater or equal to 18 years) or parental/guardian consent and patient assent (age <18 years), as required by the IRB or institution or IRB, per local regulations

Exclusion Criteria:

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients at the study site who have been treated with ClorNovir and was COVID-19 positive will be considered for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Recovery | Baseline through Day 10-End of Treatment
  Defined as the change from baseline to end of treatment in COVID-19 symptoms on a 10-item ordinal scale* ("A minimal common outcome measure set for COVID-19 clinical research," 2020).
Incidence of significant COVID-19-related clinical events | Baseline through Day 10-End of Treatment
  Such as anosmia, dysgeusia, cough, and nasal congestion.
Incidence and severity of serious adverse events (SAEs) | Baseline through Day 10-End of Treatment
Incidence and severity of adverse events (AEs) of interest | Baseline through Day 10-End of Treatment
  Such as irritation in the nasal fossa, Headache, Epistaxis, modification or discontinuation
treatment period in the incidence of hospitalizations | Baseline through Day 10-End of Treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Union Medica, Santiago de los Caballeros, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Rizvi SAA, Ferrer G, Khawaja UA, Sanchez-Gonzalez MA. Chlorpheniramine, an Old Drug with New Potential Clinical Applications: A Comprehensive Review of the Literature. Curr Rev Clin Exp Pharmacol. 2024;19(2):137-145. doi: 10.2174/2772432817666220601162006. PMID 35652393
- [Background] Taha MA, Hall CA, Shortess CJ, Rathbone RF, Barham HP. Treatment Protocol for COVID-19 Based on T2R Phenotype. Viruses. 2021 Mar 18;13(3):503. doi: 10.3390/v13030503. PMID 33803811
- [Background] Sanchez-Gonzalez, M. A., Westover, J. B., Rizvi, S. A. A., Torres, J., & Ferrer, G. A. (2022). Intranasal Chlorpheniramine Maleate for the treatment of COVID-19: Translational and Clinical Evidence. Medical Research Archives, 10(3). https://doi.org/10.18103/mra.v10i3.2752
- [Background] Torres, J., Go, C., Camacho, G., Sanchez-Gonzalez, M., & Ferrer, G. (2021). Chlorpheniramine Maleate Nasal Spray In COVID-19 Patients: Case Series. J Clin Exp Pharmacol, 10(2), 3. https://doi.org/10.35248/2161-1459.21.10.275